CLINICAL TRIAL: NCT06132438
Title: Immunotherapy Targeting of Cytomegalovirus Antigens in Glioblastoma (INTERROGATE-GBM)
Brief Title: Immunotherapy Targeting of Cytomegalovirus Antigens in Glioblastoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Charlotte Lemech (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor-Investigator, Charlotte Lemech, Principal Investigator, The University of New South Wales
Organization: The University of New South Wales (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTERROGATE-GBM
Record Dates: First submitted 2023-11-02; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glioblastoma (Experimental)
  Interventions: Drug: PEP-CMV vaccine

INTERVENTIONS:
Drug: PEP-CMV vaccine — The PEP-CMV vaccine is a long synthetic peptide (PEP) made up of 26 amino acids that is derived from the human cytomegalovirus (CMV) matrix protein pp65 and has both MHC class I and II epitopes. A vaccine platform that initially consists of TMZ-induced lymphopenia and Td pre-conditioning will be used, with serial vaccinations of up to 12 times (maximum 20) being applied. To ensure the effectiveness of the future Td pre-conditioning, which is given right before the initial PEP-CMV vaccine, a Td booster is required at enrollment.

SUMMARY:
In Australia, glioblastoma (GBM) has a higher annual fatality rate than a variety of other cancers, such as melanoma, bladder, and kidney tumors. While the 5-year survival rate for other cancers, such as breast and prostate cancer, has increased, there have been no notable advancements in GBM during the past ten years, and the incidence and mortality patterns have barely changed between 1982 and 2011. In particular, GBM poses a challenging therapeutic dilemma for patients and physicians due to its aggressive biology and resistance to available treatments. Recent studies showed that cytomegalovirus (CMV) is expressed in GBM tumors, making it a good target for immunotherapy trials. This phase I trial aims to determine the safety and tolerability of the PEP-CMV vaccine in patients with newly diagnosed MGMT-unmethylated GBM in combination with one cycle of adjuvant temozolomide.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histopathologically proven newly diagnosed primary glioblastoma.
3. Patients must have tumours which are MGMT-unmethylated.
4. Patients must be CMV-seropositive.
5. The tumour must be supratentorial.
6. Received debulking surgery. This includes complete or partial surgical resection. Biopsy alone is not acceptable.
7. Will have undergone standard concurrent radiotherapy (XRT) and temozolomide (TMZ) by the time of stage 2 participation consent.
8. Patients who are being treated with stable or decreasing doses of dexamethasone (>/= 4 mg/day) or other steroid equivalent, at the time of post-XRT adjuvant TMZ initiation.
9. Brain MRI (gadolinium-enhanced) within 31 days prior to the adjuvant TMZ.
10. Patients with neurological deficits should have deficits that are stable for a minimum of 2 weeks prior to stage 2 participant consent and should remain stable prior to the commencement of adjuvant TMZ.
11. ECOG 0-2 if >/= 70 years. ECOG 0-1 if aged > 70 years.
12. Life expectancy of > 12 weeks.
13. Adequate bone marrow function:

    * platelet count ≥ 100 x 109/L
    * absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Haemoglobin ≥ 10g/dl.
14. Adequate liver function:

    * (alanine transaminase (ALT)/aspartate transaminase (AST) ≤ 3.0 times the upper limit of normal (ULN)).
    * Total bilirubin ≤ 1.5 x ULN (Exception: Patient has known Gilbert's Syndrome or is suspected of having it, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable).
15. Adequate renal function:

    • creatinine ≤ 1.5 x ULN
16. Willing to comply with all study requirements, including treatment, timing and/or nature of required assessments
17. Signed, written informed consent.

Exclusion Criteria:

1. Pregnant or need to breastfeed during the study period (Negative serum pregnancy test required for women of childbearing potential). Not adhering to pregnancy prevention recommendations.
2. Active infection requiring treatment or an unexplained febrile (> 39 C) illness within a week of starting the trial.
3. Patients with previous inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabelled monoclonal antibodies.
4. Prior allogeneic solid organ transplant. Currently receiving or ever received immunosuppressive therapy for an organ transplant.
5. Active or prior documented autoimmune or immunosuppressive disease that has required systemic treatment (i.e. with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is allowed. Use of non-systemic topical steroids is allowed.
6. Patients receiving immunosuppressive medication or prior use within 14 days before the first dose of investigational product are excluded, except for systemic steroids up to 4 mg dexamethasone per day for the management of CNS symptoms.
7. Patients on bevacizumab or who have received prior bevacizumab as management for their GBM
8. Known human immunodeficiency virus infection and/or hepatitis B or C infections OR known to be positive for hepatitis B antigen (HBsAg)/Hepatitis B virus (HBV) DNA or Hepatitis C antibody or RNA.
9. Patients with poorly controlled, unstable or severe intercurrent medical conditions such as renal, cardiac (congestive cardiac failure, myocardial infarction within 6 months, myocarditis), or pulmonary disease or other condition, therapy or laboratory abnormality that might confound the results of the study, interfere with the patient's participation, make administration of the study drug hazardous or make it difficult to monitor adverse effects, in the opinion of the treating physician.
10. Prior conventional antitumour therapy, other than steroids, RT or TMZ therapy given for glioblastoma.
11. Allergic or unable to tolerate TMZ for any reason. Any patient that successfully completed at least 5 weeks of TMZ during standard of care XRT/TMZ and whose blood counts meet the eligibility requirements (inclusion #13) within 6 weeks post XRT/TMZ is eligible.
12. Patients receiving any other investigational drug therapy or having participated in an investigational drug/device study within 4 weeks prior to the first dose of study treatment.
13. Specific comorbidities or conditions (e.g. psychiatric) or concomitant medications which may impact the administration of study-related treatments or procedures.
14. Radiographic or cytologic evidence of leptomeningeal or multifocal disease at any time prior to treatment.
15. History of another malignancy within 2 years prior to registration. Patients with a history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or superficial transitional cell carcinoma of the bladder are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease-free for at least 2 years after definitive primary treatment.
16. Receipt of other live and attenuated vaccines within 30 days of treatment product will be excluded.
17. Unresolved toxicities from prior anticancer therapy, defined as not having resolved to NCI CTCAE grade 0 or 1, with the exception of alopecia.
18. Patients with a prior severe hypersensitivity reaction to treatment with any monoclonal antibody and/or components of the study vaccine.
19. Patients with any known severe allergies to gadolinium contrast agents.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment-related adverse events according to NCI CTCAE V5.0. | 2 weeks after the 3rd vaccine, which is approximately 12 weeks after consent.
  To assess the safety of PEP-CMV vaccination in combination with adjuvant TMZ, the percentage of patients with unacceptable toxicity will be estimated within each arm. All patients who receive any PEP-CMV vaccine will be included in these analyses.

SECONDARY OUTCOMES:
Immunologic response as measured by peak number of T cells that secrete IFNy by ELISPOT in response to component A of PEP-CMV. | Through study completion, an average of 1.5 years.